CLINICAL TRIAL: NCT06691412
Title: Obeticholic Acid Among Chronic HBV Patients with Hepatic Steatosis : Clinical and Portal Doppler Outcomes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Melad Fekry Endrawes, Assistant lecturer of internal medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: obeticholic acid in HBV
Record Dates: First submitted 2024-09-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B Virus; Steatosis
MeSH Terms: conditions — Hepatitis B; Fatty Liver | interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the group will receive obeticholic acid (Experimental): The first group that will receive obeticholic acid for six months
  Interventions: Drug: Obeticholic Acid 5 mg
- the group will not receive obeticholic acid (No Intervention): Control group

INTERVENTIONS:
Drug: Obeticholic Acid 5 mg — - Patients will be randomly divided into two groups , the first will receive obeticholic acid at a dose of 5 mg once daily and antiviral drug ,and the other will receive the antiviral drug only for six months
  Arms: the group will receive obeticholic acid

SUMMARY:
In this study, the investigators aimed to evaluate the hepatoprotective effect of OCA against HBV-induced liver injury by comparing patients demographic , laboratory date ( liver function , viremia ) , degree of hepatic steatosis and fibrosis and portal doppler at the beginning and after six months .

DETAILED DESCRIPTION:
Background :Obeticholic acid (OCA) is an agonist of the farnesoid X receptor (FXR), which plays an important role in the maintenance of bile acid homeostasis . OCA lessens liver exposure to the impact of bile acids . In addition, it binds and activates FXRs in the intestine and liver, leading to anti-inflammatory and anti-fibrotic impacts with modulation of metabolic profiles. It also inhibits the production of bile acids and increases their transport outside the hepatocytes . Activation of FXRs by OCA is 100 times higher than that exerted by chenodeoxycholic acid in attenuating intestinal and hepatic inflammation and/or fibrosis . Through modulation of bile acid homeostasis, OCA effectively reduces cholestasis-induced liver inflammation/injury.

Hepatitis B virus (HBV) is a hepatotropic virus and an important human pathogen. There are an estimated 296 million people in the world that are chronically infected by this virus, and many of them will develop severe liver diseases including hepatitis, cirrhosis and hepatocellular carcinoma (HCC).

A recent study displayed that FXR agonists potentially affect the proliferation of the hepatitis B virus (HBV). FXR agonists interact with HBV viral proteins preventing their transcription and triggering off the reduction of HBV viral protein . These findings may explain the role of OCA to antagonize HBV infection. In addition, in cirrhotic animals, OCA restored intrahepatic endothelial nitric oxide(NO) synthase levels and enhances dimethylarginine dimethylaminohydrolase 1 (DDAH1)-regulated NO production, which ultimately led to a reduction of portal pressure .

Study tools :

* All patients will be included within certain inclusion criteria after informed consent from patients and permission from the hospital board to review patients' medical records.
* Patients will be randomly divided into two groups , the first will receive obeticholic acid at a dose of 5 mg once daily and antiviral drug ,and the other will receive the antiviral drug only for six months
* All patients at the beginning of the study and at the end of six months will be subjected to:

  1. Full history taking:
* Name.
* Age.
* Sex.
* Duration of HBV infection and type of drugs 2. Anthropometric measures
* Height in cm.
* Weight in kg.
* Body mass index (kg/m²) 3. Systemic examination Including cardiac, chest and abdominal examination will be done to detect associated or excluded conditions.

  4. Laboratory tests:
  * Complete blood picture.
  * Liver function test .
  * Coagulation profile .
  * hepatitis marker (HBs Ag , Anti-HCV Ab).
  * HBV DNA PCR . 5. Radiological:
  * Fibroscan:
* The device consists of a vertically oriented mobile cuboid main body and one or several cylindrical probes. Liver stiffness measurements (LSMs) were performed after 3 hours of fasting in the right lobe of the liver through the intercostal spaces with the patient in the supine position with their right rib cage spread (which is accomplished by elevating the right hand and/or crossing the right leg over the left). After gel application, the probe is positioned perpendicular to the skin surface in one of the intercostal spaces adjacent to the right lobe of the liver (typically the 9thto 11thintercostal space, on the midaxillary line). After adequate positioning, a low frequency shear wave is induced by a small piston positioned on the tip of the probe that hits the skin surface.
* The acquired data are processed and displayed on the screen as LSM which estimate the stage of fibrosis and controlled attenuation parameter (CAP) which assess amount of steatosis.
* The examiner takes repeated measurements with the following criteria for validation:

  1. At least 10 valid measurements.
  2. Ratio of number of valid measurements to the total number of measurements is ≥ 60%.
  3. Interquartile range (IQR), which reflects the variability of measurements, is less than 30% of the median value of liver stiffness measurements .The entire exam takes approximately 5 minutes .
* CAP values range from 100 to 400 dB/m, and higher numbers indicate more pronounced steatosis. The advantage of CAP is that it is simultaneously calculated with the LSM and from the same region of interest .

CAP Score Steatosis grade Portion of liver affected by fatty change 238 to 260 dB/m S1 Less than ⅓ (11% to 33%) 260 to 290 dB/m S2 Between ⅓ and ⅔ (34% to 66%) 290 to 400 dB/m S3 More than ⅔ (67%)

- Hepatic fibrosis : LSM values range from 1.5 to 75 kPa; lower values indicate a more elastic liver. The more the liver stiffness, the more the fibrosis. The results are affected by the amount of pressure applied to the probe. The resulting LSM is translated into an estimate of the level of liver fibrosis in a simple and straightforward manner .

Liver Stiffness Result Fibrosis Score the Liver 2 to 7 kPa F0 to F1 Is normal. 8 to 9 kPa F2 Has moderate scarring. 8 to 11 kPa F3 Has severe scarring. 12 kPa or higher F4 Has cirrhosis.

* Abdominal ultrasound : to assess the liver (echogenicity, surface, edge, and size), attenuation of hepatic veins, spleen size, and presence of ascites.
* Doppler ultrasound: to measure the portal vein diameter (PVD), portal vein velocity (PVV), portal vein blood flow (PVBF), portal vein flow direction, hepatic artery resistance index and hepatic artery pulsatility index (HARI and HAPI, respectively), splenic artery resistance index (SARI), portal hypertension index (PHI), and modified liver vascular index and liver vascular index (MLVI and LVI, respectively).

Doppler analysis will be performed during quiet respiration or while the patients hold their breath . All parameters will be measured twice, at the beginning and at the end of the study. The examiner placed the Doppler gate in the hilum of the spleen and in the porta hepatis of the liver. The same observer usually will unify the method for measuring each index to avoid inter observer variability and calculate the mean of 3 consecutive measurements.

PVD : is measured from the hilar segment when crossing the inferior vena cava while the patient is in the recumbent supine position. It is recorded in millimeters.

PVBF: is calculated automatically after recording the peak, lowest, and mean venous velocity of the flow and the measurement of a cross-sectional area of the vessel lumen in a transverse plane. It is recorded in liters per minute (L/min). Portal vein flow direction: the direction of portal blood flow is shown by color Doppler, indicating if it is toward (hepatopetal) or away from the liver (hepatofugal).

PVV: is calculated automatically after measuring (Vmax) and (Vmin). It is recorded in centimeters per second (cm/sec).

HARI: The hepatic artery is evaluated by demonstrating the artery proper while crossing the portal vein. HARI is calculated automatically after measuring the hepatic artery peak velocity and end diastolic velocity measured in meters per second (m/sec) at the porta hepatis. The resistance index is calculated using the following equation: [peak systolic velocity (V max) - end diastolic velocity/peak systolic velocity (V min)/mean velocity] .

HAPI : is calculated automatically using the following equation: [(V max) - (V min)/mean velocity] .

The resistance index and wave form of the right hepatic vein: is measured as the maximum negative velocity - minimum negative velocity (or positive velocity in case of triphasic flow signal)/maximum negative velocity.

Hepatic vein waveforms : is described as triphasic, biphasic, monophasic, or not assessed because of severe attenuation.

SARI: Color Doppler allow identification of the main branches of the splenic artery by placing the transducer below the left costal margin . SARI is measured automatically after measuring (Vmax) and (Vmin), which is measured in meters per second (m/sec) by putting the cursor in the main branches of the splenic artery at the splenic hilum at the left intercostal space .

The resistance index : is calculated using the following equation: [(Vmax) - (Vmin)]/peak systolic velocity] .

PHI : is calculated as (HARI × 0.69) × (SARI × 0.87)/PVV . It is recorded in m/sec.

LVI : is calculated as PVV/HAPI . It is recorded in cm/sec. MLVI : is calculated as PVV/HARI . It is recorded in cm/sec.

5-Data management and analysis: Data collection: patients' clinical history, physical examination, laboratory results and imaging studies.

Computer software: SPSS(Statistical Package for the Social Science) version 20. Statistical tests: Data will be statistically described in terms of mean, standard deviation (SD), or frequencies (number of cases) and percentages when appropriate . A comparison of quantitative variables between the study groups will be done using Student t-test for independent samples. For comparing categorical data, Chi-square (χ2) test was performed. P values of less than 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who had diagnosed as chronic HBV on treatment with with Controlled Attenuation Parameter (CAP) value more than 238 dB/m .

Exclusion Criteria:

* patients under the age of 18.
* patients with other viral hepatitis infection .
* Hepatocellular carcinoma .
* portal vein thrombosis.
* Subjects with risk of 2nd hepatic steatosis liver disease (excessive alcohol consumption and medications).
* history of liver disease such as (α-1 antitrypsin deficiency, autoimmune hepatitis, drug-induced liver injury, 1ry biliary cirrhosis, 1ry sclerosing cholangitis).
* Body Mass Index (BMI) > 35 (to avoid the possibility of Fibroscan failure).
* Patient with end organ disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Degree of hepatic steatosis before and after six months of obeticholic acid use | 6 months
  comparing result of fibroscan regarding degree of steatosis ,controlled attenuation parameter (CAP) which assess amount of steatosis, before and after six months of using obeticholic acid

SECONDARY OUTCOMES:
portal vein doppler assesment | 6 months
  assesment of portal vein doppler before and after six months of obeticholic acid for evaluating : Portal vein flow direction and portal vein diameter : the direction of portal blood flow is shown by color Doppler, indicating if it is toward (hepatopetal) or away from the liver (hepatofugal). and the diameter is measured from the hilar segment when crossing the inferior vena cava while the patient is in the recumbent supine position. It is recorded in millimetres normal value <13 mm diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ali Mahmoud, Professor, Study Chair — Assiut University; Baha Osman Taha, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Zhang L, Duan YY, Li JM, Yin JK. Hemodynamic features of Doppler ultrasonography in patients with portal hypertension: intraoperative direct measurement of portal pressure in the portal venous system. J Ultrasound Med. 2007 Dec;26(12):1689-96. doi: 10.7863/jum.2007.26.12.1689. PMID 18029920
- [Background] Piscaglia F, Donati G, Serra C, Muratori R, Solmi L, Gaiani S, Gramantieri L, Bolondi L. Value of splanchnic Doppler ultrasound in the diagnosis of portal hypertension. Ultrasound Med Biol. 2001 Jul;27(7):893-9. doi: 10.1016/s0301-5629(01)00390-8. PMID 11476921
- [Background] Sacerdoti D, Gaiani S, Buonamico P, Merkel C, Zoli M, Bolondi L, Sabba C. Interobserver and interequipment variability of hepatic, splenic, and renal arterial Doppler resistance indices in normal subjects and patients with cirrhosis. J Hepatol. 1997 Dec;27(6):986-92. doi: 10.1016/s0168-8278(97)80141-9. PMID 9453423
- [Background] Bolognesi M, Sacerdoti D, Merkel C, Gerunda G, Maffei-Faccioli A, Angeli P, Jemmolo RM, Bombonato G, Gatta A. Splenic Doppler impedance indices: influence of different portal hemodynamic conditions. Hepatology. 1996 May;23(5):1035-40. doi: 10.1002/hep.510230515. PMID 8621130
- [Background] McNaughton DA, Abu-Yousef MM. Doppler US of the liver made simple. Radiographics. 2011 Jan-Feb;31(1):161-88. doi: 10.1148/rg.311105093. PMID 21257940
- [Background] Scheinfeld MH, Bilali A, Koenigsberg M. Understanding the spectral Doppler waveform of the hepatic veins in health and disease. Radiographics. 2009 Nov;29(7):2081-98. doi: 10.1148/rg.297095715. PMID 19926763
- [Background] Sasso M, Miette V, Sandrin L, Beaugrand M. The controlled attenuation parameter (CAP): a novel tool for the non-invasive evaluation of steatosis using Fibroscan. Clin Res Hepatol Gastroenterol. 2012 Feb;36(1):13-20. doi: 10.1016/j.clinre.2011.08.001. Epub 2011 Sep 15. PMID 21920839
- [Background] Friedrich-Rust M, Nierhoff J, Lupsor M, Sporea I, Fierbinteanu-Braticevici C, Strobel D, Takahashi H, Yoneda M, Suda T, Zeuzem S, Herrmann E. Performance of Acoustic Radiation Force Impulse imaging for the staging of liver fibrosis: a pooled meta-analysis. J Viral Hepat. 2012 Feb;19(2):e212-9. doi: 10.1111/j.1365-2893.2011.01537.x. Epub 2011 Oct 30. PMID 22239521
- [Background] Castera L, Forns X, Alberti A. Non-invasive evaluation of liver fibrosis using transient elastography. J Hepatol. 2008 May;48(5):835-47. doi: 10.1016/j.jhep.2008.02.008. Epub 2008 Feb 26. PMID 18334275
- [Background] Verbeke L, Farre R, Trebicka J, Komuta M, Roskams T, Klein S, Elst IV, Windmolders P, Vanuytsel T, Nevens F, Laleman W. Obeticholic acid, a farnesoid X receptor agonist, improves portal hypertension by two distinct pathways in cirrhotic rats. Hepatology. 2014 Jun;59(6):2286-98. doi: 10.1002/hep.26939. Epub 2014 Apr 14. PMID 24259407
- [Background] Erken R, Andre P, Roy E, Kootstra N, Barzic N, Girma H, Laveille C, Radreau-Pierini P, Darteil R, Vonderscher J, Scalfaro P, Tangkijvanich P, Flisiak R, Reesink H. Farnesoid X receptor agonist for the treatment of chronic hepatitis B: A safety study. J Viral Hepat. 2021 Dec;28(12):1690-1698. doi: 10.1111/jvh.13608. Epub 2021 Sep 29. PMID 34467593
- [Background] GBD 2019 Hepatitis B Collaborators. Global, regional, and national burden of hepatitis B, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Gastroenterol Hepatol. 2022 Sep;7(9):796-829. doi: 10.1016/S2468-1253(22)00124-8. Epub 2022 Jun 21. PMID 35738290
- [Background] Fiorucci S, Di Giorgio C, Distrutti E. Obeticholic Acid: An Update of Its Pharmacological Activities in Liver Disorders. Handb Exp Pharmacol. 2019;256:283-295. doi: 10.1007/164_2019_227. PMID 31201552
- [Background] Chapman RW, Lynch KD. Obeticholic acid-a new therapy in PBC and NASH. Br Med Bull. 2020 May 15;133(1):95-104. doi: 10.1093/bmb/ldaa006. PMID 32282030
- [Background] Nevens F, Andreone P, Mazzella G, Strasser SI, Bowlus C, Invernizzi P, Drenth JP, Pockros PJ, Regula J, Beuers U, Trauner M, Jones DE, Floreani A, Hohenester S, Luketic V, Shiffman M, van Erpecum KJ, Vargas V, Vincent C, Hirschfield GM, Shah H, Hansen B, Lindor KD, Marschall HU, Kowdley KV, Hooshmand-Rad R, Marmon T, Sheeron S, Pencek R, MacConell L, Pruzanski M, Shapiro D; POISE Study Group. A Placebo-Controlled Trial of Obeticholic Acid in Primary Biliary Cholangitis. N Engl J Med. 2016 Aug 18;375(7):631-43. doi: 10.1056/NEJMoa1509840. PMID 27532829
- [Background] Cao P, Gan J, Wu S, Hu Y, Xia B, Li X, Zeng H, Cheng B, Yu H, Li F, Si L, Huang J. Molecular mechanisms of hepatoprotective effect of tectorigenin against ANIT-induced cholestatic liver injury: Role of FXR and Nrf2 pathways. Food Chem Toxicol. 2023 Aug;178:113914. doi: 10.1016/j.fct.2023.113914. Epub 2023 Jun 20. PMID 37348807